CLINICAL TRIAL: NCT06578949
Title: A Phase 3, Single-arm, Open-label, Multicenter Study to Assess the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Ravulizumab in Complement Inhibitor Treatment Naïve Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) in China
Brief Title: Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Ravulizumab in Chinese Adults Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9289C00008; ALXN1210-PNH-323 (Other: Alexion)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; Ravulizumab
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): During the Primary Treatment Period, participants will receive a weight-based loading dose of ravulizumab on Day 1 followed by weight-based maintenance dose of ravulizumab on Day 15 and once every 8 weeks (q8w) thereafter for a total of 26 weeks. On Day 183, all participants will enter a 32-week Extension Treatment Period and receive ravulizumab. Beginning on Day 183, participants will receive a maintenance dose of ravulizumab q8w for an additional 32 weeks.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Ravulizumab will be administered by intravenous (IV) infusion.
  Other Names: ALXN1210

SUMMARY:
The primary objective of this study is to evaluate the efficacy of ravulizumab in adult participants with PNH.

ELIGIBILITY:
Inclusion Criteria:

* Adult C5 inhibitor naive PNH patients (age>=18), which is confirmed by flow cytometry evaluation.
* Must be vaccinated againast N meningitidis.

Exclusion Criteria

* Meningitidis infection or unresolved meningococcal disease
* History of bone marrow transplantation
* Other significant systemic diseases that might have impact on efficacy and safety assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Lactate Dehydrogenase (LDH) From Baseline to Day 183 (Week 26) | Baseline, Day 183 (Week 26)

SECONDARY OUTCOMES:
Number of Participants Achieving LDH <1.5 × Upper Limit of Normal (ULN) at Day 183 (Week 26) | Day 183 (Week 26)
Number of Participants Achieving Transfusion Avoidance (TA) Through Day 183 (Week 26) | Day 183 (Week 26)
Number of Participants Experiencing Breakthrough Hemolysis Through Day 183 (Week 26) | Day 183 (Week 26)
Change in Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) Score From Baseline to Day 183 (Week 26) | Day 183 (Week 26)
Change in Hemoglobin (Hgb) From Baseline to Day 183 (Week 26) | Baseline, Day 183 (Week 26)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nantong
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR